CLINICAL TRIAL: NCT02274480
Title: Diffusion Weighted Imaging as a Biomarker for Detection of Chemotherapy Induced Cardiotoxicity
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-191
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Chemotherapy Induced Cardiotoxicity in Breast Cancer Patients
Keywords: MRI; Diffusion Weighted Imaging; 14-191
MeSH Terms: interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Breast cancer patients with cardiotoxicity: Each patient will undergo a cardiac MRI with DWI. The standard of care in patients with declining LVEF is a cardiac MRI. For this study, those patients will also have the added DWI sequence. For patients who are not already scheduled for a cardiac MRI by their referring physician, and therefore do not have an upcoming standard of care cardiac MRI, a research cardiac MRI with DWI will be added. They will not be charged for the DW-MRI of the heart or any additional images taken as part of that scan. Patients unable to tolerate lying flat for this length of time or to tolerate the scan for any reason will be withdrawn and replaced in the study. After their cardiac MRI, their participation in the study is complete.
  Interventions: Device: cardiac MRI with DWI
- Breast cancer patients without cardiotoxicity: Each patient will undergo a cardiac MRI with DWI. The standard of care in patients with declining LVEF is a cardiac MRI. For this study, those patients will also have the added DWI sequence. For patients who are not already scheduled for a cardiac MRI by their referring physician, and therefore do not have an upcoming standard of care cardiac MRI, a research cardiac MRI with DWI will be added. They will not be charged for the DW-MRI of the heart or any additional images taken as part of that scan. Patients unable to tolerate lying flat for this length of time or to tolerate the scan for any reason will be withdrawn and replaced in the study. After their cardiac MRI, their participation in the study is complete.
  Interventions: Device: cardiac MRI with DWI

INTERVENTIONS:
Device: cardiac MRI with DWI

SUMMARY:
The goal of this study is to see if a special type of heart scan called a diffusion weighted magnetic resonance imaging (DW-MRI) that uses extra measurements, can be used to find early signs of heart damage from chemotherapy.

DETAILED DESCRIPTION:
This prospective single institutional pilot study will enroll breast cancer patients who develop cardiotoxicity while on anthracycline and anti-HER2 therapy . The control group will be composed of patients on similar anthracycline therapy and dose but without a decline in LVEF on Cardiac MRI (CMR). Clinic visits with monitoring for cardiotoxicity occur as part of standard of care after therapy initiation. The study and control group will be composed of 15 patients each. At the discretion of the treating physician, patients will be recruited from the Breast Medical Oncology Service.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age on the day of signing the informed consent.
* Diagnosis of HER2+ breast cancer

  * History of anthracycline therapy and antiHER2 treatment
* For subjects with decrease in LVEF: Recent (within 12 weeks) drop in LVEF ≥10% on echocardiogram from baseline and confirmed by cardiac MRI for the study population. If the drop in EF is not confirmed on MRI, the subject will be removed and placed into the control group.

For control group: Less than a 10% change in EF from baseline for the control population confirmed on echocardiogram and cardiac MRI. If no change in EF is not confirmed on MRI, the subject will be removed and placed into the study group if the change in EF is equal to or greater than 10%. Note: Male breast cancer patients are uncommon and are not expected to be included in this study, however if they meet the above criteria, they will not be excluded.

Exclusion Criteria:

* Prior myocardial infarction
* Prior surgical or percutaneous coronary revascularization
* Pregnant or lactating patients
* Patients who because of general medical or psychiatric condition, or physiologic status unrelated to the presence of breast cancer cannot give valid informed consent
* Patients who are unwilling or unable to undergo MRI including patients with contraindications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips, claustrophobia, inability to lie flat for the duration of the study etc. MRI eligibility will be determined on the day of consent with the MRI questionnaire.
* Patients with metallic implants or device in the chest that might distort local magnetic field and compromise quality of MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the selection criteria will be recruited from the breast medical oncology clinics at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
presence of edema | 1 year
  associated with cardiotoxicity as visualized on DWI by the attending cardiac imagers we may explore the association of the presence of edema on DWI with a drop in LVEF > 10% using exact logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Plodkowski, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/